CLINICAL TRIAL: NCT07195838
Title: Effects of a Hybrid, Personalised Mindfulness-optimised Pulmonary Rehabilitation (Mindful-Breath) Programme for Active Living for People With Chronic Obstructive Pulmonary Disease: A Pilot Randomised Controlled Trial
Brief Title: Mindful-Breath for People With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Kwok Yan Yan, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22233241
Record Dates: First submitted 2025-06-23; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Mindfulness; Pulmonary Rehabilitation; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: mindfulness; pulmonary rehabilitation; chronic obstructive pulmonary disease; RCT; lifestyle modification; mHealth; EMI; physical inactivity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: hybrid mindfulness-based pulmonary rehabilitation and lifestyle modification group (Experimental): (i) Eight 60-min hybrid group sessions, combining mindfulness-based pulmonary rehabilitation and lifestyle modification. The sessions cover topics such as the eight yoga's ethical guidelines (yamas and niyamas) for positive lifestyle behaviors, breathing mechanisms, dysfunctional breathing styles, voluntary control of breathing (pranayama), relaxation and sense withdrawal (pratyahara), concentration (dharana), meditation (dhyana), and enlightenment (samadhi). Subsequent sessions will be delivered via videoconferencing using Zoom and will include guided breathing-focused practices.
  (ii) Ecological Momentary Interventions (EMI):Personalised mindfulness-based lifestyle counselling through instant messages with chat-based support throughout the 8-week intervention period.
  (iii) Activity Monitoring: All participants will wear a wristband activity tracker to monitor their physical activity in daily life.
  Interventions: Behavioral: Hybrid Mindfulness-Based Group Sessions; Behavioral: Ecological Momentary Interventions (EMI); Device: Activity Monitoring
- Control: Single General Education on Pulmonary Rehabilitation and Lifestyle Modification Group (Active Comparator): (i) The control group participants will receive a single in-person 60-min group session on general education on pulmonary rehabilitation and lifestyle modification based on the GOLD 2024 teaching set and HEARTS technical package for NCD prevention as recommended by the WHO, and will only receive reminder messages for follow-ups. (ii) Activity Monitoring: All participants will wear a wristband activity tracker to monitor their physical activity in daily life.
  Interventions: Behavioral: Single General Education on Pulmonary Rehabilitation and Lifestyle Modification Group; Device: Activity Monitoring

INTERVENTIONS:
Behavioral: Hybrid Mindfulness-Based Group Sessions — Eight 60-min hybrid group sessions, combining mindfulness-based pulmonary rehabilitation and lifestyle modification. The sessions cover topics such as the eight yoga's ethical guidelines (yamas and niyamas) for positive lifestyle behaviors, breathing mechanisms, dysfunctional breathing styles, voluntary control of breathing (pranayama), relaxation and sense withdrawal (pratyahara), concentration (dharana), meditation (dhyana), and enlightenment (samadhi). Subsequent sessions will be delivered via videoconferencing using Zoom and will include guided breathing-focused practices.
  Arms: Intervention: hybrid mindfulness-based pulmonary rehabilitation and lifestyle modification group
Behavioral: Ecological Momentary Interventions (EMI) — Personalised mindfulness-based lifestyle counselling through instant messages with chat-based support throughout the 8-week intervention period. The intervention protocol will cover message content library, regular message delivery and personalised chat-based support.
  Arms: Intervention: hybrid mindfulness-based pulmonary rehabilitation and lifestyle modification group
Behavioral: Single General Education on Pulmonary Rehabilitation and Lifestyle Modification Group — The control group participants will receive a single in-person 60-min group session on general education on pulmonary rehabilitation and lifestyle modification based on the GOLD 2024 teaching set and HEARTS technical package for NCD prevention as recommended by the WHO.
  Arms: Control: Single General Education on Pulmonary Rehabilitation and Lifestyle Modification Group
Device: Activity Monitoring — All participants will wear a wristband activity tracker to monitor their physical activity in daily life.

SUMMARY:
Individuals living with chronic obstructive pulmonary disease (COPD) often suffer from stress and behavioral risks such as physical inactivity. In an attempt to promote healthy behaviors and overall wellbeing among this particular population, this study aims to develop and evaluate a personalized Mindful-Breath intervention combining telehealth technology and mindfulness for COPD patients. This is an assessor-blinded, two-arm exploratory randomized controlled trial with a sequential mixed-method design. A total of 60 participants will be recruited and randomly assigned to either intervention or control group using 1:1 ratio. Intervention group will go through 8 weekly 60-min hybrid group sessions, combining mindfulness-based pulmonary rehabilitation and lifestyle modification. Personalized mindfulness-based lifestyle counselling through instant messages with chat-based support throughout the 8-week intervention period will also be provided. Control group will receive a single in-person 60-min group session on general education on pulmonary rehabilitation and lifestyle modification and will only receive reminder messages for follow-ups. Variables such as time spent on physical activity, lung function, perceived stress, symptom burden and health-related quality of life will be collected at three time-points (T0: baseline, prior to randomization; T1: immediate post-intervention; T2: 3-month post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-80 years
* Sex: Male or female
* Education level: Primary or above
* Diagnosis: COPD (Baseline FEV1 <80% and FEV1/FVC <70% of predicted normal values)
* Severity of COPD: Stage I to IV
* Group of COPD: Group B, or E, based on 2024 GOLD guideline (36)
* Clinical stability: No acute exacerbation in the past 4 weeks. Patients with recent acute exacerbation in the past 4 weeks will be screened again in subsequent follow-up.
* Moderate stress: PSS score ≥14 (28)
* Access to a mobile device (e.g., a smartphone, tablet, or laptop) with internet connectivity
* Ability to read, communicate, and provide written consent in Chinese.

Exclusion Criteria:

* Engaging in >60 minutes/week of moderate PA based on American Lung Association guidelines
* Recent or ongoing receipt of other pharmacological/behavioral trials within the past 3 months
* Contraindications or severe comorbidities that may limit full participation (mental diseases, deafness, limb activity disorder, coronary heart disease, arterial aneurysm, uncontrolled hypertension, pregnancy, etc)
* Co-existing respiratory diseases (Asthma/interstitial lung disease/bronchiectasis) or active malignancies
* Very severe COPD requiring long-term oxygen therapy or home non-invasive ventilation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility in terms of rates of recruitment, retention and adherence | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention)
  The feasibility of interventions will be evaluated in terms of rates of recruitment, retention, and adherence. Reasons for these rates will be recorded.
Acceptability in terms of instances of adverse events | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention)
  Instances of adverse events (information regarding physical and psychological problems will be kept)
Acceptability in terms of satisfaction with intervention | T1 (immediate post-intervention)
  Satisfaction with intervention will be measured by a questionnaire rating on four key domains: usefulness of treatment, opinion of the therapist, perceived improvement and likelihood to recommend the treatment to others

SECONDARY OUTCOMES:
Time spent on moderate-vigorous PA in the past week (min) | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention)
  Time spent on moderate-vigorous PA in the past week (min) measured by a smartwatch. The data will be considered valid if the participants wear the smartwatch for ≥10 hours/days for ≥5 days in the past week of assessment time-point
Self-reported PA in the past week | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Self-reported PA in the past week will be measured by the validated 9-item International Physical Activity Questionnaire Short-form (IPAQ-SF)(Chinese), which records four intensity PA levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Pulmonary function | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Pulmonary function will be evaluated using portable spirometry. The assessment includes measuring forced expiratory volume in 1s (FEV1), forced vital capacity (FVC), peak expiratory flow (PEF), and oxygen saturation (SaO2). The highest value for FEV1, FVC, and EFV1/FVC (Tiffeneau-Pinelli index) from three reproducible efforts will be recorded.
Perceived stress | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Perceived stress will be measured by the validated 10-item Perceived Stress Scale (PSS)(Chinese)(Cronbach's α: 0.78-0.91). The event frequency of each item in the last month will be rated using a five-point Likert scale. Higher scores indicate higher perceived stress levels.
Spiritual well-being | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Spiritual well-being measured by the validated Chinese Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being 12-Item Scale (FACIT-Sp-12), which assess three constructs: belief, meaning and sense of peace on a 4-point Likert scale. High scores indicate high levels of spiritual well-being.
Symptom burden and HRQOL | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Symptom burden and HRQOL will be measured by the validated disease-specific 50-item St. George's Respiratory Questionnaire (SGRQ)(Chinese), which assesses three domains: frequency and severity of respiratory symptoms, effects of breathlessness on mobility and PA, and psychosocial impact of the disease. Scores are weighted such that every domain score and the total score range from 0-100. Higher scores indicate a poorer HRQOL. The minimally clinically important response to treatment is defined as an improvement of 4% on the separate domains and the total score.
Impact of COPD on daily life | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Impact of COPD on daily life will be measured by the COPD Assessment Test (CAT). This patient-completed questionnaire evaluates the overall effect of COPD-specifically symptoms such as cough, sputum, dyspnea, and chest tightness-on health status. CAT scores range from 0 to 40, with higher scores indicating a more severe impact of COPD on a patient's life. A five-unit difference in scores distinguishes stable patients from those experiencing exacerbations.
Breathlessness | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Breathlessness will be measured by the modified Medical Research Council (mMRC) Dyspnoea scale. The mMRC scale is a self-assessment tool used to measure the level of impairment caused by breathlessness during daily activities, rated on a scale from 0 (no breathlessness except on strenuous exercise) to 4 (too breathless to leave the house, or breathless when dressing or undressing).
Cardiopulmonary functions | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Cardiopulmonary functions will be assessed through the 6-minute walk test, where distance walked, oxygen saturation (SpO2), and heart rate will be measured.
Exacerbation in the follow-up period | Repeated outcome measures will be collected at three time-points (T0:baseline, prior to randomisation; T1: immediate post-intervention; T2: 3-month post-intervention).
  Exacerbation in the follow-up period will be recorded to better to understand the frequency and severity of COPD exacerbations, contributing to a comprehensive understanding of disease management and progression.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are available upon request from the principal investigator, Prof. Kwok. These data are not publicly available, as they contain information that could compromise the privacy of research participants.